CLINICAL TRIAL: NCT00159978
Title: Validation of 18F-MISO-PET and 18F-FLT-PET by Immunohistochemical Assessment of Head and Neck Cancer Resection Specimen
Brief Title: Validation of 18F-MISO-PET and 18F-FLT-PET
Status: Terminated | Type: Observational
Why Stopped: Problems with FMISO supply
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 100
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Head and Neck Neoplasms
Keywords: head and neck cancer; hypoxia; tumor cell proliferation; PET
MeSH Terms: conditions — Head and Neck Neoplasms; Hypoxia | interventions — alovudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor resection specimen
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: 18F-FLT and 18F-MISO-PET — 18F-FLT-PET-images will be acquired one hour after injection of 250 MBq FLT. 18F-MISO-PET: 400 MBq FMISO will be injected intravenously. Marker administration: The day before surgery (≤ 24h) pimonidazole (500 mg/m2) will be administered intravenously in 100 ml saline over 20 min. IdUrd (200 mg) will be administered as bolus injection 20 min before surgery.

SUMMARY:
Hypoxia and tumor cell proliferation are important mechanisms contributing to resistance to radiotherapy in human head and neck tumor cells. Currently, assessment of these two tumor characteristics is performed in biopsies using immunohistochemical staining and subsequent analysis. A promising non-invasive method of characterizing a tumor is the use of positron-emission tomography (PET). Specific tracers can be used to detect hypoxia and proliferative activity. 18F-misonidazole is a tracer for hypoxia and 18F-thymidine is a tracer for proliferation.

Patients suffering from head and neck cancer and who will undergo surgery will be included in this study.

One week before the surgery the patients will undergo a CT-scan and a PET-scan with either of the tracers. Shortly before the surgery they will be given immunohistochemically detectable marker substances enabling the characterization of the tumor samples gathered from the resection specimen. These markers are pimonidazole for detection of hypoxia and iododeoxyuridine for detection of tumor cell proliferation.

The data collected by PET-scan will be analysed and compared to the results acquired by immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Stage II-IV squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx, planned for curative resection.
* Age >18 years.
* Written informed consent.

Exclusion Criteria:

* Pregnancy.
* Prior treatment for this tumor
* Women breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Squamous cell carcinoma of the head and neck
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2005-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To validate 18F-MISO-PET for detection of tumor hypoxia and 18F-FLT-PET for detection of tumor cell proliferation by immunohistochemical assessment of hypoxia and proliferation in head and neck cancer resection specimen. | 1 month

SECONDARY OUTCOMES:
To assess if functional information obtained by 18F-MISO-PET and 18F-FLT-PET can improve the definition of target volume for radiotherapy treatment planning. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Johannes HA Kaanders, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- UMC St Radboud, Department of Radiotherapy, Nijmegen, Gelderland, Netherlands